CLINICAL TRIAL: NCT00195975
Title: Heart Rate Variability in Children With Abdominal Pain Related to a Functional Gastrointestinal Disorder: Relationship to Anxiety/Stress, Electrogastrography, and Rapid Water Loading
Brief Title: Heart Rate Variability in Children With a Functional Gastrointestinal Disorder
Status: Completed | Type: Observational
Sponsor: Children's Mercy Hospital Kansas City (Other)
Responsible Party: Jennifer Verrill Schurman, Ph.D./Principal Investigator, Children's Mercy Hospital
Other Study IDs: 00005085
Record Dates: First submitted 2005-09-14; First posted 2005-09-20 (Estimated); Last update posted 2011-06-28 (Estimated); Status verified 2011-06

CONDITIONS: Abdominal Pain
Keywords: Abdominal Pain; Functional Gastrointestinal Disorders; Stress; Anxiety; Autonomic Nervous System
MeSH Terms: conditions — Abdominal Pain; Gastrointestinal Diseases; Anxiety Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: Children with FD
- 4: Healthy controls

SUMMARY:
The current study is designed to assess relationships between anxiety/stress, autonomic nervous system balance, and electrical activity in the stomach before and after eating/drinking in children with abdominal pain.

DETAILED DESCRIPTION:
Chronic or recurrent abdominal pain in children is a very common complaint in children and adolescents, and is most often associated with the presence of a functional gastrointestinal disorder (FGID). It is likely that the clinical symptoms in FGIDs are the result of an interaction between biologic, psychologic, and social factors. The psychologic factor most implicated is chronic stress or anxiety. Stress may influence gastrointestinal function and symptoms through altering the balance of the autonomic nervous system (ANS). Imbalance in the ANS has potential effects on gastrointestinal mechanosensitivity, motor function (e.g. stomach emptying and accommodation), and electrical rhythms. All of these can be associated with abdominal pain. Theory and early evidence from studies done with healthy adult populations suggest that ANS imbalance can reduce the body's ability to respond electrically to food/water consumption. However, the relationships between chronic stress/anxiety, ANS balance/imbalance, and electrical activity in the stomach before and after eating/drinking remain to be fully explored in children with FGIDs. The current study is a two-part pilot study designed to assess these relationships. Part I involves assessment of anxiety/stress (i.e., BASC parent- and self-reports) along with ANS balance (i.e., heart rate variability) and electrical activity in the stomach (i.e., electrogastrography) measured in the fasting state and following a test meal. Part II involves the same assessments with rapid water loading replacing the test meal. Results will be analyzed by specific FGID, as well as for the group as a whole. We expect to enroll 75 children ages 8-17 in each part, including 30 healthy controls and 45 children with an FGID. Elucidating these relationships is a necessary first step in developing more effective treatments for children with recurrent abdominal pain and, ultimately, reducing the personal and societal costs of this common pain entity.

ELIGIBILITY:
Inclusion Criteria:

* Ages 8 - 17 years
* Evaluated in Abdominal Pain Clinic at Children's Mercy Hospital or the Gastroenterology Clinic at Children's Mercy South for abdominal pain of at least 8 weeks duration and fulfilling symptom-based criteria for FD, IBS, or FD/IBS.

Exclusion Criteria:

* Previous abdominal surgery
* Chronic disease requiring regular medical care (e.g. gastrointestinal diseases, diabetes mellitus, juvenile rheumatoid arthritis, cystic fibrosis, cancer).
* Non-English speaking

NOTE: Control subjects will meet all patient inclusion/exclusion criteria except for Inclusion Criteria #2. Control subjects will be excluded for history of abdominal pain, nausea, vomiting, diarrhea, constipation, or bloating.

Ages: 8 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children with IBS, FD, or IBS and FD, as well as healthy controls without these conditions.
Sampling Method: Non-Probability Sample
Enrollment: 44 (Actual)
Dates: Start 2005-06; Primary Completion 2008-08 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
HRV or the magnitude of power in the LF or HF in the fasting or post-prandial state | Same day
HRV or stress profile parameters following an acute stress(mental math) | Same day
Frequency of an abnormal EGG or the magnitude of EGG parameters | Same day
Water load volume | Same day

SECONDARY OUTCOMES:
Behavioral Assessment System for Children (BASC) | Same day
Salivary cortisol | Same day
A stress profile via the biofeedback equipment (e.g. measures of muscle tension, hand temperature, and skin moisture (conductance). | Same day

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer V Schurman, PhD, Principal Investigator — Children's Mercy Hospital Kansas City
Locations (1):
- Children's Mercy Hospital and Clinics, Kansas City, Missouri, United States